CLINICAL TRIAL: NCT04901312
Title: Identifying an Effective and Cost Beneficial Approach to Preventing OUD in Justice-Involved Youth
Brief Title: Preventing OUD in Justice-Involved Youth
Acronym: POST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other); Washington State Department of Children, Youth and Families (Unknown); Michigan State University (Other); RTI International (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kym Ahrens, Associate Professor, Division of Adolescent Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-131-DCYF; UG3DA050189 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-05-25 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Substance Use Disorders; Recidivism
Keywords: Juvenile Rehabilitation; Adolescent; Young Adult; Juvenile Justice; Opioids; Opioid Use Disorder; Substance Use; Prevention; Recidivism; Substance Use Disorder; Cost Effectiveness; Benefit Cost Analysis
MeSH Terms: conditions — Substance-Related Disorders; Recidivism; Opioid-Related Disorders | interventions — Educational Status; Therapeutics; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial
Who Masked: Outcomes Assessor
Masking Description: The Outcomes Assessor (data collection team) will not be aware of the participant's study arm when they collect survey data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced A-CRA (E-ACRA) (Experimental): Higher intensity
  Interventions: Behavioral: Adolescent Community Reinforcement Approach; Behavioral: Assertive Continuing Care; Behavioral: Trauma Affect Regulation Guide for Education and Therapy; Behavioral: Motivational Interviewing; Other: Opioid Education Workbook
- Assertive Community Support (ACS) (Experimental): Lower intensity
  Interventions: Behavioral: Adolescent Community Reinforcement Approach; Behavioral: Assertive Continuing Care; Behavioral: Motivational Interviewing; Other: Opioid Education Workbook

INTERVENTIONS:
Behavioral: Adolescent Community Reinforcement Approach — The Adolescent Community Reinforcement Approach (A-CRA) is a developmentally-appropriate behavioral treatment for youth and young adults ages 12 to 24 years old with substance use disorders. A-CRA seeks to increase the family, social, and educational/vocational reinforces to support recovery. This intervention has been implemented in outpatient, intensive outpatient, and residential treatment settings. A-CRA includes guidelines for three types of sessions: individuals alone, parents/caregivers alone, and individuals and parents/caregivers together. According to the individual's needs and self-assessment of happiness in multiple life areas, clinicians choose from a variety of A-CRA procedures that address, for example, problem-solving skills to cope with day-to-day stressors, communication skills, and active participation in positive social and recreational activities with the goal of improving life satisfaction and eliminating alcohol and substance use problems.
  Other Names: A-CRA; ACRA
Behavioral: Assertive Continuing Care — Assertive Continuing Care (ACC) uses Community Reinforcement Approach (CRA) procedures, home visits, and case management for individuals following an initial substance use treatment episode. It stresses rapid initiation of services after discharge from residential, intensive outpatient, or regular outpatient treatment in order to promote recovery and prevent relapse.
  Other Names: ACC
Behavioral: Trauma Affect Regulation Guide for Education and Therapy — Trauma Affect Regulation: Guide for Education and Therapy is a psychosocial intervention for traumatized adolescents, adults, and families, and for workforce and organizational responses to secondary/vicarious traumatization. T4, the 4-session version, provides education about the impact of complex traumatic stress on the brain's stress response system, and strengths-based practical skills for re-setting the trauma-related alarm/survival reactions that occur in complex PTSD.
  Other Names: T4; TARGET
  Arms: Enhanced A-CRA (E-ACRA)
Behavioral: Motivational Interviewing — Motivational interviewing is a collaborative, person-centered form of guiding to elicit and strengthen motivation for change.
  Other Names: MI
Other: Opioid Education Workbook — A digital workbook designed to be completed on a computer in about 2 hours. Topics include opioid use, opioid use disorder, and prevention and treatment of opioid overdose.
  Other Names: Education

SUMMARY:
The United States is experiencing an opioid epidemic. Sadly, opioid-related fatalities are on the rise, causing profound emotional, financial, and cultural impacts. One way to reduce these negative impacts is to prevent people from developing opioid use problems in the first place.

Research shows that youth and young adults in the juvenile justice system have higher rates of opioid use disorder than other young people in the general population. The POST Study seeks develop, implement and evaluate the effectiveness and cost of 2 opioid use prevention programs of varying intensities. The prevention programs are designed specifically for youth and young adults living in justice settings. It is implemented during the time they are transitioning out of incarceration and back into the community. The research team hopes their results will help justice settings implement their own effective opioid prevention programs in the future.

DETAILED DESCRIPTION:
Non-prescription opioid use in adolescents and young adults is epidemic in our country and overdose-related fatalities are rising. Adolescents and young adults in justice settings have some of the highest rates of opioid use disorder (OUD), with national rates approaching 20%. The majority of these youth and young adults engage in problematic non-opioid substance use, which is a critical risk factor for OUD. Non-opioid substance use disorders (SUDs) and OUD, in turn, are two of the most important predictors of subsequent re-involvement in juvenile or criminal justice systems.

In this study, researchers at Seattle Children's Research Institute, the University of Washington, Michigan State University, and Washington State Juvenile Rehabilitation/Department of Children Youth and Families will collaboratively develop and test an evaluation of OUD prevention interventions of varying intensities based on the Adolescent Community Reinforcement Approach with Assertive Continuing Care (ACRA+ACC). Multiple studies have established effectiveness of ACRA+ACC in reducing SUD; however, none has evaluated it as an OUD prevention strategy. SUD is incredibly common and costly among youth and young adults involved in juvenile justice systems.

Thus, ACRA+ACC-based approaches are likely to be effective and cost-beneficial OUD prevention strategies for this group.

Investigators seek to determine the optimal intensity of an ACRA+ACC-based OUD prevention intervention for AYAJS with and without non-opioid SUD, as these groups are likely to have differing prevention needs. To do so, they will use a Sequential Multiple Assignment Randomized Trial (SMART) study design to construct high-quality adaptive interventions with ACRA+ACC-based OUD prevention strategies of different intensity levels among youth with and without SUD. Based on self-reported substance use at 1 month post-release, participants may be re-randomized into another study arm. This will both address treatment need and provide data for subsequent effectiveness and cost analyses.

In Phase I of this study, researchers collaboratively planned for a SMART experiment, i.e.: finalize infrastructure, recruitment, intervention, and data collection procedures; and create infrastructure for the possibility of future implementation of effective interventions. They conducted a pilot with 31 participants to assess feasibility of protocols and procedures, recruitment, engagement, and retention strategies in anticipation of a future larger trial. Phase I started in January 2021.

In Phase II of this study, currently ongoing, researchers are conducting a SMART trial with 215 AYAJS aged 15-25, with or without SUD but without moderate or severe OUD, to evaluate ACRA/ACC-based interventions of various intensity levels for youth. They will also conduct cost, cost-effectiveness, and benefit-cost analyses to understand the relationships between intervention costs and outcomes. Phase II started in August 2021.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-25
* Leaving a Washington State detention facility or group home in the next 5-7 months
* Able to speak/understand English sufficiently to participate meaningfully in the intervention and assessments

Exclusion Criteria:

* Diagnosed with a moderate or severe Opioid Use Disorder
* Has a learning or mental health issue severe enough that they are unable to participate meaningfully in the intervention and assessments (e.g. schizophrenia or severe developmental disability)

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 215 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of substance use episodes | Last 30 days at 2 months post-release (Phase I)
  Self-reported number of episodes of substance use on days any substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of substance use episodes | Last 30 days at 3 months post-release (Phase II)
  Self-reported number of episodes of substance use on days any substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of substance use episodes | Last 30 days at 6 months post-release (Phase II)
  Self-reported number of episodes of substance use on days any substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Frequency of substance use episodes | Last 30 days at 2 months post-release (Phase I)
  Self-reported number of days of any substance use in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Frequency of substance use episodes | Last 30 days at 3 months post-release (Phase II)
  Self-reported number of days of any substance use in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Frequency of substance use episodes | Last 30 days at 6 months post-release (Phase II)
  Self-reported number of days of any substance use in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Rate of Recidivism | 12 months post-release
  Convictions in either the juvenile or adult justice system for offenses within an 18-month period
Rate of Recidivism | 18 months post-release
  Convictions in either the juvenile or adult justice system for offenses within an 18-month period

SECONDARY OUTCOMES:
Number of new opioid users | 6 months post-release (Phase II)
  Number of participants who ever used opioids among those who had never used at baseline based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of participants with escalated opioid use | Last 30 days at 2 months post-release vs. before incarceration (Phase I)
  Number of participants whose days of use increased compared to prior measure based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of participants with escalated opioid use | Last 30 days at 3 months post-release vs. before incarceration (Phase II)
  Number of participants whose days of use increased compared to prior measure based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of participants with escalated opioid use | Last 30 days at 6 months post-release vs. at 3 months post-release (Phase II)
  Number of participants whose days of use increased compared to prior measure based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of use episodes of specific substances (e.g. opioids, marijuana, etc.) | Last 30 days at 2 months post-release (Phase I)
  Self-reported number of episodes of use of a specific substance on days that substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of use episodes of specific substances (e.g. opioids, marijuana, etc.) | Last 30 days at 3 months post-release (Phase II)
  Self-reported number of episodes of use of a specific substance on days that substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of use episodes of specific substances (e.g. opioids, marijuana, etc.) | Last 30 days at 6 months post-release (Phase II)
  Self-reported number of episodes of use of a specific substance on days that substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Frequency of use of specific substances (e.g. opioids, marijuana, etc.) | Last 30 days at 2 months post-release (Phase I)
  Self-reported number of days a specific substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Frequency of use of specific substances (e.g. opioids, marijuana, etc.) | Last 30 days at 3 months post-release (Phase II)
  Self-reported number of days a specific substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Frequency of use of specific substances (e.g. opioids, marijuana, etc.) | Last 30 days at 6 months post-release (Phase II)
  Self-reported number of days a specific substance was used in the past 30 days based on questions developed in collaboration with coordinating center Research Triangle Institute and other grantees.
Number of instances of overdose among non-opioid users | Last 30 days at 3 months post-release (Phase II)
  Self-reported number of instances of overdose
Number of instances of overdose among non-opioid users | Last 30 days at 6 months post-release (Phase II)
  Self-reported number of instances of overdose
Problematic substance use | Last 30 days at 6 months post-release (Phase II)
  Self-reported substance use beyond a developmentally appropriate threshhold. For those under age 21, problematic use is defined as any of the following: 1) use of alcohol or marijuana several times a week or more; 2) use of any other drugs, or dabbing marijuana 1-2 times per month or more; 3) score on CRAFFT of 2 or more (https://crafft.org).
  For those age 21 and older, problematic use is defined as any of the following: 1) use of alcohol or marijuana every day or most days each week; 2) use of any other drugs, or dabbing marijuana 1-2 times per month or more; 3) score on CRAFFT of 2 or more (https://crafft.org)
Problematic substance use | Last 30 days at 3 months post-release (Phase II)
  Self-reported substance use beyond a developmentally appropriate threshhold. For those under age 21, problematic use is defined as any of the following: 1) use of alcohol or marijuana several times a week or more; 2) use of any other drugs, or dabbing marijuana 1-2 times per month or more; 3) score on CRAFFT of 2 or more (https://crafft.org).
  For those age 21 and older, problematic use is defined as any of the following: 1) Use of alcohol or marijuana every day or most days each week; 2) Use of any other drugs, or dabbing marijuana 1-2 times per month or more; 3) Score on CRAFFT of 2 or more (https://crafft.org)
Cost of ACRA Lite (medium intensity arm) per participant | 3 months post-release
  Cost in US Dollars of ACRA Lite intervention from study's Cost Analysis program
Cost of Enhanced ACRA (high intensity arm) per participant | 3 months post-release
  Cost in US Dollars of Enhanced ACRA intervention from study's Cost Analysis program
Cost of Education Workbook (low intensity arm) per participant | at release
  Cost in US Dollars of Education Workbook intervention from study's Cost Analysis program

OTHER OUTCOMES:
Participant attendance | 2 months post-release (Phase I)
  Number of sessions attended
Participant attendance | 3 months post-release (Phase II)
  Number of sessions attended
Participant satisfaction | 2 months post-release (Phase I)
  Self-reported satisfaction with coach on a scale of very satisfied, somewhat satisfied, not very satisfied, not at all satisfied
Participant satisfaction | 3 months post-release (Phase II)
  Self-reported satisfaction with coach on a scale of very satisfied, somewhat satisfied, not very satisfied, not at all satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Kym Ahrens, MD MPH, Principal Investigator — Seattle Children's Hospital; Kevin Haggerty, MSW PhD, Principal Investigator — University of Washington
Locations (1):
- Washington State Department of Children, Youth and Families, Olympia, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with other researchers in the HEAL Prevention Collaborative. Further specific detail will be reported as the plans are finalized.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Within four weeks of acceptance by a journal, we will deposit electronic copies of publications in PubMed Central.
  Publications will be made publicly available immediately without any embargo period.

REFERENCES:
- [Background] Martins SS, Segura LE, Santaella-Tenorio J, Perlmutter A, Fenton MC, Cerda M, Keyes KM, Ghandour LA, Storr CL, Hasin DS. Prescription opioid use disorder and heroin use among 12-34 year-olds in the United States from 2002 to 2014. Addict Behav. 2017 Feb;65:236-241. doi: 10.1016/j.addbeh.2016.08.033. Epub 2016 Aug 30. No abstract available. PMID 27614657
- [Background] Understanding the epidemic. Retrieved from https://www.cdc.gov/drugoverdose/epidemic/index.html. Accessed 3-2-2019.2018.
- [Background] Forsyth CJ, Biggar RW, Chen J, Burstein K. Examining heroin use and prescription opioid misuse among adolescents. Criminal Justice Studies: A Critical Journal of Crime, Law & Society 2017;30:320-9.
- [Background] Sung HE, Richter L, Vaughan R, Johnson PB, Thom B. Nonmedical use of prescription opioids among teenagers in the United States: trends and correlates. J Adolesc Health. 2005 Jul;37(1):44-51. doi: 10.1016/j.jadohealth.2005.02.013. PMID 15963906
- [Background] Vaughn MG, Fu Q, Perron BE, Wu LT. Risk profiles among adolescent nonmedical opioid users in the United States. Addict Behav. 2012 Aug;37(8):974-7. doi: 10.1016/j.addbeh.2012.03.015. Epub 2012 Mar 27. PMID 22525786
- [Background] Wojciechowski TW. Developmental Trajectories of Opioid Use Among Juvenile Offenders: An Epidemiological Examination of Group Characteristics and Criminological Risk Factors. Subst Use Misuse. 2019;54(7):1203-1213. doi: 10.1080/10826084.2019.1573837. Epub 2019 Feb 15. PMID 30767596
- [Background] Mulvey EP, Schubert CA, Chassin L. Substance Use and Offending in Serious Adolescent Offenders. In: Department of Justice OoJP, Office of Juvenile Justice and Delinquency Prevention., ed. Washington, DC: U.S. 2010.
- [Background] Grisso T. Double jeopardy: adolescent offenders with mental disorders. Chicago: University of Chicago Press; 2004.
- [Background] Ghandour LA, El Sayed DS, Martins SS. Alcohol and illegal drug use behaviors and prescription opioids use: how do nonmedical and medical users compare, and does motive to use really matter? Eur Addict Res. 2013;19(4):202-10. doi: 10.1159/000345445. Epub 2013 Feb 7. PMID 23391856
- [Background] Cheng T, Small W, Nosova E, Hogg B, Hayashi K, Kerr T, DeBeck K. Nonmedical prescription opioid use and illegal drug use: initiation trajectory and related risks among people who use illegal drugs in Vancouver, Canada. BMC Res Notes. 2018 Jan 16;11(1):35. doi: 10.1186/s13104-018-3152-9. PMID 29338770
- [Background] Jones CM, McCance-Katz EF. Co-occurring substance use and mental disorders among adults with opioid use disorder. Drug Alcohol Depend. 2019 Apr 1;197:78-82. doi: 10.1016/j.drugalcdep.2018.12.030. Epub 2019 Feb 14. PMID 30784952
- [Background] Scott T, Brown SL. Risks, strengths, gender, and recidivism among justice-involved youth: A meta-analysis. J Consult Clin Psychol. 2018 Nov;86(11):931-945. doi: 10.1037/ccp0000343. PMID 30335425
- [Background] The National Center for Addiction and Substance Abuse Research, Columbia University. Criminal Neglect: Substance Abuse, Juvenile Justice and The Children Left Behind. 2004.
- [Background] Mulvey EP. Highlights From Pathways to Desistance: A Longitudinal Study of Serious Adolescent Offenders. 2011.
- [Background] Godley SH, Smith JE, Meyers RJ, Godley MD. The Adolescent Community Reinforcement Approach: A Clinical Guide for Treating Substance Use Disorders. Normal, IL: Chestnut Health Systems; 2016.
- [Background] Godley SH, Meyers RJ, Smith JE, et al. The Adolescent Community Reinforcement Approach for Adolescent Cannabis Users (Cannabis Youth Treatment (Cyt) Series) - Volume 4. Rockville, MD.
- [Background] Ahrens KR, Dubois DL, Garrison M, Spencer R, Richardson LP, Lozano P. Qualitative exporation of relationships with important non-parental adults in the lives of youth in foster care. Child Youth Serv Rev. 2011 Jun 1;33(6):1012-1023. doi: 10.1016/j.childyouth.2011.01.006. PMID 22661797
- [Background] Godley MD, Passetti LL, Subramaniam GA, Funk RR, Smith JE, Meyers RJ. Adolescent Community Reinforcement Approach implementation and treatment outcomes for youth with opioid problem use. Drug Alcohol Depend. 2017 May 1;174:9-16. doi: 10.1016/j.drugalcdep.2016.12.029. Epub 2017 Feb 22. PMID 28282523
- [Background] Godley SH, Hedges K, Hunter B. Gender and racial differences in treatment process and outcome among participants in the adolescent community reinforcement approach. Psychol Addict Behav. 2011 Mar;25(1):143-54. doi: 10.1037/a0022179. PMID 21443309
- [Background] Godley SH, Hunter BD, Fernandez-Artamendi S, Smith JE, Meyers RJ, Godley MD. A comparison of treatment outcomes for adolescent community reinforcement approach participants with and without co-occurring problems. J Subst Abuse Treat. 2014 Apr;46(4):463-71. doi: 10.1016/j.jsat.2013.10.013. Epub 2013 Nov 11. PMID 24462478
- [Background] Henderson CE, Wevodau AL, Henderson SE, Colbourn SL, Gharagozloo L, North LW, Lotts VA. An independent replication of the Adolescent-Community Reinforcement Approach with justice-involved youth. Am J Addict. 2016 Apr;25(3):233-40. doi: 10.1111/ajad.12366. Epub 2016 Mar 18. PMID 26992083
- [Background] Meyers RJ, Roozen HG, Smith JE. The community reinforcement approach: an update of the evidence. Alcohol Res Health. 2011;33(4):380-8. PMID 23580022
- [Background] Fleming C, Haggerty K. Process and Outcomes Evaluation of Keys to Success. 2013.
- [Background] Almirall D, Nahum-Shani I, Sherwood NE, Murphy SA. Introduction to SMART designs for the development of adaptive interventions: with application to weight loss research. Transl Behav Med. 2014 Sep;4(3):260-74. doi: 10.1007/s13142-014-0265-0. PMID 25264466
- [Background] Florence CS, Zhou C, Luo F, Xu L. The Economic Burden of Prescription Opioid Overdose, Abuse, and Dependence in the United States, 2013. Med Care. 2016 Oct;54(10):901-6. doi: 10.1097/MLR.0000000000000625. PMID 27623005
- [Background] Pain in the nation: The drug, alcohol and suicide crises and the need for a national resilience strategy. 2017. (Accessed September 25, 2018, at http://www.paininthenation.org/assets/pdfs/TFAH-2017- PainNationRpt.pdf.)
- [Background] Centers for Disease Control and Prevention (CDC). CDC grand rounds: prescription drug overdoses - a U.S. epidemic. MMWR Morb Mortal Wkly Rep. 2012 Jan 13;61(1):10-3. PMID 22237030
- [Background] Opioids. 2016. (at https://www.samhsa.gov/atod/opioids.)
- [Background] Case A, Deaton A. Mortality and morbidity in the 21st century. Brookings Pap Econ Act. 2017 Spring;2017:397-476. doi: 10.1353/eca.2017.0005. PMID 29033460
- [Background] Opioid epidemic. 2016. (Accessed September 25, 2018, at https://www.atg.wa.gov/opioid-epidemic.)
- [Background] Schulenberg JE, Johnston LD, O'Malley PM, Bachman JG, Miech RA, Patrick ME. Monitoring the Future national survey results on drug use, 1975-2017: Volume II, College students and adults ages 19-55. Ann Arbor: Institute for Social Research, The University of Michigan; 2018.
- [Background] Jones CM. Heroin use and heroin use risk behaviors among nonmedical users of prescription opioid pain relievers - United States, 2002-2004 and 2008-2010. Drug Alcohol Depend. 2013 Sep 1;132(1-2):95-100. doi: 10.1016/j.drugalcdep.2013.01.007. Epub 2013 Feb 12. PMID 23410617
- [Background] Banerjee G, Edelman EJ, Barry DT, Becker WC, Cerda M, Crystal S, Gaither JR, Gordon AJ, Gordon KS, Kerns RD, Martins SS, Fiellin DA, Marshall BD. Non-medical use of prescription opioids is associated with heroin initiation among US veterans: a prospective cohort study. Addiction. 2016 Nov;111(11):2021-2031. doi: 10.1111/add.13491. Epub 2016 Aug 23. PMID 27552496
- [Background] Charak R, Ford JD, Modrowski CA, Kerig PK. Polyvictimization, Emotion Dysregulation, Symptoms of Posttraumatic Stress Disorder, and Behavioral Health Problems among Justice-Involved Youth: a Latent Class Analysis. J Abnorm Child Psychol. 2019 Feb;47(2):287-298. doi: 10.1007/s10802-018-0431-9. PMID 29654539
- [Background] Perez NM, Jennings WG, Baglivio MT. A path to serious, violent, chronic delinquency: The harmful aftermath of adverse childhood experiences. Crime & Delinquency 2018;64:3-25.
- [Background] Abbott PJ. A review of the community reinforcement approach in the treatment of opioid dependence. J Psychoactive Drugs. 2009 Dec;41(4):379-85. doi: 10.1080/02791072.2009.10399776. PMID 20235445
- [Background] Roozen HG, Boulogne JJ, van Tulder MW, van den Brink W, De Jong CA, Kerkhof AJ. A systematic review of the effectiveness of the community reinforcement approach in alcohol, cocaine and opioid addiction. Drug Alcohol Depend. 2004 Apr 9;74(1):1-13. doi: 10.1016/j.drugalcdep.2003.12.006. PMID 15072802
- [Background] Carroll KM, Ball SA, Nich C, Martino S, Frankforter TL, Farentinos C, Kunkel LE, Mikulich-Gilbertson SK, Morgenstern J, Obert JL, Polcin D, Snead N, Woody GE; National Institute on Drug Abuse Clinical Trials Network. Motivational interviewing to improve treatment engagement and outcome in individuals seeking treatment for substance abuse: a multisite effectiveness study. Drug Alcohol Depend. 2006 Feb 28;81(3):301-12. doi: 10.1016/j.drugalcdep.2005.08.002. Epub 2005 Sep 28. PMID 16169159
- [Background] Goossens I, Nicholls TL, Torchalla I, Brink J, de Ruiter C. The Perceived Impact of Trauma-Focused Research on Forensic Psychiatric Patients With Lifetime Victimization Histories. J Empir Res Hum Res Ethics. 2016 Oct;11(4):334-345. doi: 10.1177/1556264616670769. Epub 2016 Nov 25. PMID 27887006
- [Background] Catalano RF, Park J, Harachi TW, Haggerty KP, Abbott RD, Hawkins JD. Mediating the effects of poverty, gender, individual characteristics, and external constraints on antisocial behavior: A test of the social development model and implications for developmental life-course theory. In: Farrington DP, ed. Advances in criminological theory: Vol 14. New Brunswick, NJ: Transaction; 2005:99-123.
- [Background] Catalano RF, Hawkins JD. The social development model: A theory of antisocial behavior. In: Hawkins JD, ed. Delinquency and crime: Current theories. New York: Cambridge University Press; 1996:149-97.
- [Background] Hirschi T. Causes of delinquency. Berkeley, CA: University of California Press; 1969.
- [Background] Bandura A. Social learning theory. Englewood Cliffs, NJ: Prentice Hall; 1977.
- [Background] Sutherland EH. Development of the theory [Private paper published posthumously]. In: Schuessler K, ed. Edwin Sutherland on analyzing crime. Chicago: University of Chicago Press; 1973:13-29.
- [Background] R.L. M. The current state of differential association theory. Crime and Delinquency 1988;34:277-306.
- [Background] Catalano RF, Gainey RR, Fleming CB, Haggerty KP, Johnson NO. An experimental intervention with families of substance abusers: one-year follow-up of the focus on families project. Addiction. 1999 Feb;94(2):241-54. doi: 10.1046/j.1360-0443.1999.9422418.x. PMID 10396792
- [Background] Fleming CB, Catalano RF, Oxford ML, Harachi TW. A test of generalizability of the social development model across gender and income groups with longitudinal data from the elementary school developmental period. Journal of Quantitative Criminology 2002;18:423-39.
- [Background] Ford JD, Grasso DJ, Greene CA, Slivinsky M, DeViva JC. Randomized clinical trial pilot study of prolonged exposure versus present centred affect regulation therapy for PTSD and anger problems with male military combat veterans. Clin Psychol Psychother. 2018 Sep;25(5):641-649. doi: 10.1002/cpp.2194. Epub 2018 Apr 23. PMID 29687524
- [Background] Ford JD, Chang R, Levine J, Zhang W. Randomized clinical trial comparing affect regulation and supportive group therapies for victimization-related PTSD with incarcerated women. Behav Ther. 2013 Jun;44(2):262-76. doi: 10.1016/j.beth.2012.10.003. Epub 2012 Nov 5. PMID 23611076
- [Background] Ford JD, Grasso DJ, Hawke J, Chapman JF. Poly-victimization among juvenile justice-involved youths. Child Abuse Negl. 2013 Oct;37(10):788-800. doi: 10.1016/j.chiabu.2013.01.005. Epub 2013 Feb 19. PMID 23428165
- [Background] Ford JD, Steinberg KL, Hawke J, Levine J, Zhang W. Randomized trial comparison of emotion regulation and relational psychotherapies for PTSD with girls involved in delinquency. J Clin Child Adolesc Psychol. 2012;41(1):27-37. doi: 10.1080/15374416.2012.632343. PMID 22233243
- [Background] Ford JD, Steinberg KL, Zhang W. A randomized clinical trial comparing affect regulation and social problem-solving psychotherapies for mothers with victimization-related PTSD. Behav Ther. 2011 Dec;42(4):560-78. doi: 10.1016/j.beth.2010.12.005. Epub 2011 Apr 16. PMID 22035986
- [Background] www.wsipp.wa.gov/BenefitCost?topicId=1 Accessed 3-2-2019.
- [Derived] Kuklinski MR, Gibbons BJ, Bowser DM, McCollister KE, Smart R, Dunlap LJ, Shenkar E, Bonar EE, Boomer T, Campbell M, Fiellin LE, Hutton DW, Rao V, Saldana L, Su K, Walton MA, Yilmazer T. Investing in Interventions to Prevent Opioid Use Disorder in Adolescents and Young Adults: Start-up Costs from NIDA's HEAL Prevention Initiative. Prev Sci. 2025 Nov;26(7):1045-1055. doi: 10.1007/s11121-025-01835-6. Epub 2025 Oct 14. PMID 41085955
- [Derived] Brincks AM, Haggerty KP, Kolberg A, Albertson KM, McCarty CA, Kuklinski MR, Ryle T, Ahrens KR. Development of the Positive Outcomes through Supported Transition (POST) opioid preventive intervention for youth in the legal system: Study protocol for a sequential multiple assignment randomized trial. Contemp Clin Trials. 2025 Feb;149:107782. doi: 10.1016/j.cct.2024.107782. Epub 2024 Dec 18. PMID 39706330
- [Derived] Ahrens KR, Brincks AM, Haggerty KP, McCarty CA, Dean S, Albertson KM, Cross SR, Ryle T, Wun A. Designing and piloting a sequential multiple assignment randomized trial for opioid prevention among youth in the legal system. Psychol Addict Behav. 2025 Feb;39(1):14-26. doi: 10.1037/adb0001025. Epub 2024 Sep 9. PMID 39250243
- [Derived] Ahrens K, Blackburn N, Aalsma M, Haggerty K, Kelleher K, Knight DK, Joseph E, Mulford C, Ryle T, Tolou-Shams M. Prevention of Opioid Use and Disorder Among Youth Involved in the Legal System: Innovation and Implementation of Four Studies Funded by the NIDA HEAL Initiative. Prev Sci. 2023 Oct;24(Suppl 1):99-110. doi: 10.1007/s11121-023-01566-6. Epub 2023 Jul 1. PMID 37393415
- See also: Mortality and morbidity in the 21st century — https://www.brookings.edu/bpea-articles/mortality-and-morbidity-in-the-21st-century.)
- See also: The opioid epidemic — https://www.atg.wa.gov/opioid-epidemic
- See also: Benefit-Cost Analysis — http://www.wsipp.wa.gov/BenefitCost?topicId=1